CLINICAL TRIAL: NCT00002909
Title: A PHASE I CLINICAL AND PHARMACOLOGIC EVALUATION OF PHENYLBUTYRATE IN PATIENTS WITH REFRACTORY SOLID TUMORS: STUDY OF CONTINUOUS EXPOSURE ORAL PHENYLBUTYRATE ON A THREE TIMES DAILY SCHEDULE
Brief Title: Phenylbutyrate in Treating Patients With Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02250; J-9616; JHOC-9616; NCI-T95-0017H; CDR0000065274 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2001-02

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Drug Therapy; 4-phenylbutyric acid

ARMS (1):
- Arm I (Experimental): All patients receive oral phenylbutyrate three times daily. Groups of 4 or more patients receive escalating doses of phenylbutyrate until the maximum tolerated dose (MTD) is determined. Treatment continues until disease progression or unacceptable toxicity intervenes.
  Interventions: Drug: chemotherapy; Drug: oral sodium phenylbutyrate

INTERVENTIONS:
Drug: chemotherapy
Drug: oral sodium phenylbutyrate

SUMMARY:
Phase I trial to study the effectivenes of phenylbutyrate in treating adults with refractory solid tumor or lymphoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of oral phenylbutyrate that can be given three times daily in patients with refractory solid tumors or lymphoma until disease progression or a trough plasma concentration of 2-6 micromoles per liter is achieved.

II. Characterize the pharmacokinetics of oral phenylbutyrate absorption, and determine whether there is time dependence in the systemic clearance rate during multiple dosing.

III. Seek preliminary evidence of therapeutic activity of phenylbutyrate when administered on this schedule in these patients.

IV. Correlate any observed responses and toxic effects with results of bioassays and tissue sampling for phenylbutyrate activity.

OUTLINE: This is a dose-seeking study.

All patients receive oral phenylbutyrate three times daily. Groups of 4 or more patients receive escalating doses of phenylbutyrate until the maximum tolerated dose (MTD) is determined. Treatment continues until disease progression or unacceptable toxicity intervenes.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor or lymphoma that is progressive or refractory to conventional therapy or for which no effective therapy is known
* Priority given to hormone-refractory prostate cancer and melanoma
* No untreated CNS metastases
* Head CT not required in the absence of clinical signs or symptoms but recommended for metastatic melanoma

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-2
* Life expectancy: At least 3 months
* WBC greater than 2,000/mm3 OR absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin greater than 9 g/dL
* Bilirubin less than 1.5 mg/dL
* AST/ALT less than 1.5 times normal
* Creatinine less than 2.0 mg/dL
* Obstructive uropathy allowed if relieved by nephrostomy or other appropriate device
* Left ventricular ejection fraction greater than 40% by MUGA or normal by echocardiogram
* No history of congestive heart failure
* No uncontrolled hypertension (diastolic greater than 110 mm Hg)
* Forced expiratory volume (1 second) greater than 1.5 L/min
* No active infection, including HIV or viral hepatitis
* No active seizure disorder
* No clinical evidence of increased intracranial pressure
* No baseline dementia (mini-mental exam less than 23)
* No autoimmune disease, including systemic lupus erythematosus, scleroderma, or other connective tissue illness
* No nonmalignant medical or psychiatric problem of sufficient severity to limit full compliance with study or to pose undue risk
* Not pregnant or nursing
* Adequate contraception required of fertile patients for 2 weeks prior to, during, and for 3 months after study
* Normal gastrointestinal function with ability to tolerate large intake of oral volume required for phenylbutyrate administration
* Patients with persistent nausea or moderate to severe anorexia may not be good candidates for study

PRIOR CONCURRENT THERAPY:

* Fully recovered from all prior therapy
* Prior suramin allowed if serum suramin level less than 50 micrograms/mL at entry
* At least 28 days since chemotherapy
* No prior phenylacetate, phenylbutyrate, or antineoplaston therapy
* The following may be continued during study:
* Luteinizing hormone-releasing hormone agonist with evidence of tumor progression (e.g., rising prostate-specific antigen, new lesions on bone scan) despite therapy
* Adrenal steroid replacement (if needed)
* Dexamethasone or other steroids
* At least 4-6 weeks since flutamide with evidence of PSA progression required (if possible)
* At least 28 days since radiotherapy
* At least 28 days since major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1997-02; Primary Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Carducci, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States

REFERENCES:
- [Result] Carducci M, Bowling MK, Eisenberger M, et al.: Phenylbytyrate (PB) for refractory solid tumors: Phase I evaluation of continuous oral PB exposure. [Abstract] Proc Am Assoc Cancer Res 39: A507, 1998.